CLINICAL TRIAL: NCT01357642
Title: Epinephrine Inhalation Aerosol USP, an HFA-MDI: Clinical Study-C For Evaluation Of Efficacy And Safety In Asthma Patients
Brief Title: Epinephrine Inhalation Aerosol USP: For Evaluation Of Efficacy And Safety In Asthma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: API-E004-CL-C
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Asthma
Keywords: asthma; bronchial asthma; shortness of breath
MeSH Terms: conditions — Asthma; Dyspnea | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm T (Experimental): Arm T is the experimental treatment arm consisting of 2 x 125 mcg/inhalations of E004, QID, with 4-6 hr intervals
  Interventions: Drug: Epinephrine inhalation aerosol
- Arm P (Placebo Comparator): Placebo comparator as 2×Placebo QID, with 4-6 hr intervals
  Interventions: Drug: Placebo
- Arm A (Active Comparator): Active comparator, Primatene Mist, 2×220 mcg/inhalation, QID, with 4-6 hr intervals
  Interventions: Drug: epinephrine inhalation aerosol

INTERVENTIONS:
Drug: Epinephrine inhalation aerosol — Epinephrine inhalation aerosol, 125 mcg/inhalation, 2 inhalations QID at 4 - 6 hour intervals
  Other Names: epinephrine inhalation aerosol - HFA propelled
  Arms: Arm T
Drug: Placebo — Placebo for epinephrine inhalation aerosol, formulation without epinephrine
  Arms: Arm P
Drug: epinephrine inhalation aerosol — epinephrine inhalation aerosol, 220 mcg/inhalation, 2 inhalations QID at 4-6 hour intervals
  Other Names: Primatene Mist
  Arms: Arm A

SUMMARY:
This clinical study evaluates the 12-week efficacy and safety of Epinephrine HFA Inhalation Aerosol HFA the proposed HFA formulation of metered dose inhaler (MDI) of Epinephrine, in comparison to a Placebo-HFA control MDI and the currently marketed Primatene® Mist (epinephrine CFC inhaler), in adolescent and adult subjects with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented asthma, requiring inhaled epinephrine or beta 2-agonist treatment.
* No significant changes in asthma therapy and no asthma-related hospitalization or emergency visits, within 4 weeks prior to Screening
* Can tolerate withholding treatment with inhaled bronchodilators and other allowed medications for the minimum washout period.
* Demonstrating a Screening Baseline FEV1 that is 50 - 90% of predicted normal value.
* Demonstrating at least a 12% Airway Reversibility.
* Demonstrating satisfactory techniques in the use of metered-dose inhaler and a hand held peak expiratory flow meter.
* Female patients of child-bearing potential must be non-pregnant and non-lactating at Screening and throughout the study, and must use an acceptable method of contraception during the study.

Exclusion Criteria:

* A smoking history of 10-pack years, or having smoked within 12 months of screening.
* Any current or past medical conditions that, per investigator discretion, might significantly affect responses to the study drugs, other than asthma.
* Concurrent clinically significant diseases.
* Known intolerance or hypersensitivity to any component of the study drugs.
* Recent infection of the respiratory tract, before screening.
* Use of prohibited medications.
* Having been on other investigational drug/device studies in the last 30 days prior to screening.
* Known or highly suspected substance abuse.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in Area Under the Curve (AUC) versus placebo | at 5, 30, 60, 120, 180, 240, and 360 minutes post-dose
  Serial FEV1 measurements to demonstrate the mean AUC of change in percent FEV1 from same-day baseline of E004 (Treatment T; Epinephrine-HFA) versus Placebo-HFA (Treatment P) is the primary efficacy endpoint.

SECONDARY OUTCOMES:
Monitor vital signs | 2, 10, 20, 60, and 360 min after dosing
  Assess blood pressure, pulse rate
Cardiac rhythm | at baseline, 2, 10, 20, and 60 min post-dose
  At study visits 1 and 5 only, perform 12 lead ECG
Blood glucose and potassium | baseline, and at 15 and 120 min post-dose
  Monitor blood glucose and potassium levels to assure appropriate balance

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - West Coast Clinical Trials, Costa Mesa, California
  - Southern California Institute for Respiratory Diseases, Los Angeles, California
  - Asthma and Allergy Associates of Southern California, Mission Viejo, California
  - CHOC PSF, Division of Allergy, Asthma and Immunology, Orange, California
  - Allergy & Asthma Assocaites of Santa Clara Valley, San Jose, California
  - Colorado Allergy & Asthma Centers, Centennial, Colorado
  - Colorado Allergy & Asthma Centers, Denver, Colorado
  - Rocky Mountain Center for Clinical Research, Wheat Ridge, Colorado
  - Atlanta Allergy & Asthma Clinic, Woodstock, Georgia
  - Iowa Clinical Research Corporation, Iowa City, Iowa
  - Family Allergy & Asthma Research Institute, Louisville, Kentucky
  - Northeast Medical Research Associates, No. Dartmouth, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - Clinical Research Institute, Plymouth, Minnesota
  - The Clinical Research Center, St Louis, Missouri
  - Clinical Research Group of Montana, Bozeman, Montana
  - The Asthma & Allergy Center, Bellevue, Nebraska
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - North Carolina Clinical Research, Raleigh, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Intergated Medical Research, Ashland, Oregon
  - Allergy and Asthma Research Group, Eugene, Oregon
  - Baker Allergy, Asthma & Dermatology Research Center, Lake Oswego, Oregon
  - The Clinical Research Institute of Southern Oregon, Medford, Oregon
  - Transitional Clinical Research, Portland, Oregon
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Asthma & Allergy Research Associates, Upland, Pennsylvania
  - National Allergy, Asthma & Urticaria Centers of Charleston, Charleston, South Carolina
  - Western Sky Research, El Paso, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy Partners, Richmond, Virginia
  - ASTHMA, Inc., Seattle, Washington

REFERENCES:
- [Background] Pinnas JL, Schachtel BP, Chen TM, Roseberry HR, Thoden WR. Inhaled epinephrine and oral theophylline-ephedrine in the treatment of asthma. J Clin Pharmacol. 1991 Mar;31(3):243-7. doi: 10.1002/j.1552-4604.1991.tb04969.x. PMID 2019665
- [Background] Hendeles L, Marshik PL, Ahrens R, Kifle Y, Shuster J. Response to nonprescription epinephrine inhaler during nocturnal asthma. Ann Allergy Asthma Immunol. 2005 Dec;95(6):530-4. doi: 10.1016/S1081-1206(10)61014-9. PMID 16400891
- [Background] Warren JB, Doble N, Dalton N, Ewan PW. Systemic absorption of inhaled epinephrine. Clin Pharmacol Ther. 1986 Dec;40(6):673-8. doi: 10.1038/clpt.1986.243. PMID 3780129
- [Background] Cripps A, Riebe M, Schulze M, Woodhouse R. Pharmaceutical transition to non-CFC pressurized metered dose inhalers. Respir Med. 2000 Jun;94 Suppl B:S3-9. PMID 10919679
- [Background] Dickinson BD, Altman RD, Deitchman SD, Champion HC. Safety of over-the-counter inhalers for asthma: report of the council on scientific affairs. Chest. 2000 Aug;118(2):522-6. doi: 10.1378/chest.118.2.522. PMID 10936150
- [Background] Simons FE, Gu X, Johnston LM, Simons KJ. Can epinephrine inhalations be substituted for epinephrine injection in children at risk for systemic anaphylaxis? Pediatrics. 2000 Nov;106(5):1040-4. doi: 10.1542/peds.106.5.1040. PMID 11061773
- [Derived] Kerwin EM, Tashkin DP, Korenblat PE, Greos LS, Pearlman DS, Bensch GW, Miller SD, Marrs T, Luo MZ, Zhang JY. Long-term safety and efficacy studies of epinephrine HFA metered-dose inhaler (Primatene(R) Mist): a two-stage randomized controlled trial. J Asthma. 2021 May;58(5):633-644. doi: 10.1080/02770903.2020.1713147. Epub 2020 Jan 20. PMID 31959019